CLINICAL TRIAL: NCT04309669
Title: Assessment of the eFficacy, the Onset-of-Action and the Safety of Tot'héma® in Adults With Moderate Iron Deficiency Anaemia
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoire Innotech International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOT401-19
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tot'hema (Experimental): three ampoules per day during 12 weeks daily dose: 150mg of iron per day.
  Interventions: Drug: TOT'HEMA

INTERVENTIONS:
Drug: TOT'HEMA — three ampoules per day during 12 weeks

SUMMARY:
The aim of this study is to assess, in patients with moderate IDA, the Onset-of-Action of a daily treatment with Tot'Héma®. The onset of action is defined as the time required for a mean increase of at least 0,5g/dL from baseline in the haemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women (>18 years)
2. Patient with a confirmation of moderate anemia defined as: 8 g/dL ≤ Haemoglobin level ≤ 9 g/dL on the last hematological test performed within 7 days before inclusion visit.
3. Patient with ferritin blood level < lower limit of laboratory standard for this biological parameter at on the last hematological test performed within 7 days before inclusion visit.
4. Patient who has read, understood, dated and signed the informed consent form

6. Patient agreeing to comply with protocol requirements, including visits and blood samples at specifically defined dates

Non-inclusion Criteria:

1. Patient for whose an oral iron supplementation is not indicated or not recommended according to PI's opinion
2. CRP > 10 mg/L on the last hematological test performed within 7 days before inclusion visit.
3. Patient with benign or malignant neoplastic tumour
4. Patient presenting gastrointestinal disorders incompatible with study treatment compliance
5. Pregnant or breastfeeding woman
6. Woman with childbearing potential who does not agree to use an accepted highly effective method of contraception - per investigator's judgment
7. Patient with surgery scheduled to occur during the treatment period
8. Patient allergic or hypersensitive to any of the components of Tot'Héma® ampoule
9. Patient with chronic inflammatory disease, including chronic inflammatory bowel syndrome and/or chronic heart failure and/or chronic renal failure and/or inflammatory rheumatism
10. Patient with active digestive bleeding (such as digestive ulcer)
11. Patient having taken iron supplementation, iron-based IV therapy or mineral supplementation with iron, within the 15 days prior to the inclusion visit (V2)
12. Patient with fructose intolerance, glucose-galactose malabsorption syndrome or sucrase-isomaltase deficiency
13. Patient with acute malaria crisis within 15 days prior to inclusion
14. Patient with a positive Faecal Occult Blood Test (FOBT)
15. Patient with HIV infection
16. Unreliable patients, including non-observant patients, patients with known alcoholism or drug abuse, or with a history of a serious psychiatric disorder, as well as patients who are reluctant to give informed consent or to comply with protocol requirement.

Selection criterion 1. Patient with moderate anaemia defined as 8 g/dL ≤ haemoglobin level ≤ 9 g/dL on the last hematological test performed within 7 days before screening visit

Inclusion criteria

1. Adult men and women (≥18 years) 2. Patient with a confirmation of moderate anaemia defined as 8 g/dL ≤ haemoglobin level ≤ 9 g/dL on the last hematological test performed within 7 days before inclusion visit 3. Patient with ferritin blood level < lower limit of laboratory standard for this biological parameter on the last hematological test performed within 7 days before inclusion visit 4. Patient who has read, understood, dated and signed the informed consent form 5. Patient agreeing to comply with protocol requirements, including visits and blood samples at specifically defined dates Non-inclusion criteria

1. Patient for whom an oral iron supplementation is not indicated or not recommended according to Investigator's opinion
2. C-Reactive Protein > 10 mg/L on the last hematological test performed within 7 days before inclusion visit
3. Patient with benign or malignant neoplastic tumour
4. Patient presenting gastrointestinal disorders incompatible with study treatment compliance
5. Pregnant or breastfeeding woman
6. Woman with childbearing potential who does not agree to use an accepted highly effective method of contraception - per investigator's judgment
7. Patient with surgery scheduled to occur during the treatment period
8. Patient allergic or hypersensitive to any of the components of Tot'héma® ampoule
9. Patient with chronic inflammatory disease, including chronic inflammatory bowel syndrome and/or chronic heart failure and/or chronic renal failure and/or inflammatory rheumatism
10. Patient with active digestive bleeding (such as digestive ulcer)
11. Patient having taken iron supplementation, iron-based IV therapy mineral supplementation with iron within the 15 days prior to the inclusion visit (V2)
12. Patient with fructose intolerance, glucose-galactose malabsorption syndrome or sucrase-isomaltase deficiency
13. Patient with acute malaria crisis within 15 days prior to inclusion
14. Patient with a positive Faecal Occult Blood Test (FOBT)
15. Patient with HIV infection
16. Unreliable patients, including non-observant patients, patients with known alcoholism or drug abuse, or with a history of a serious psychiatric disorder, as well as patients who are reluctant to give informed consent or to comply with protocol requirement.
17. Patient with a family relationship to a person at the investigator's site or at the Sponsor or at the CRO.
18. Participant involved in another interventional or observational clinical trial or who participated in another interventional clinical trial within four weeks before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Time required for a mean increase of at least 0,5g/dL from baseline in the haemoglobin level in patients with moderate IDA and daily treated with Tot'héma. | 12 weeks
  Identification of the first time (in days) associated with a mean increase in the haemoglobin level of at least 0.5 g/dL (versus mean haemoglobin level at D0).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitié Salpétrière - Médecine Interne et Immunologie Clinique, Paris, France

REFERENCES:
- [Derived] Cacoub P, Otieno FO, Trichereau J, Gobert O, Kerveillant AL, Escola J, Verriere F. Early Haematologic Response to Oral Iron Treatment in Adults With Moderate Iron-Deficiency Anaemia. Anemia. 2025 Nov 20;2025:8866390. doi: 10.1155/anem/8866390. eCollection 2025. PMID 41277915